CLINICAL TRIAL: NCT00379236
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of EUFLEXXA™ for Treatment of Painful Osteoarthritis of the Knee, With an Open-Label Safety Extension
Brief Title: A Study of the Efficacy and Safety of EUFLEXXA™ for Treatment of Painful Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-01D
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Results first posted 2009-12-10 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EUFLEXXA™ Double-blind (Experimental): Each subject received 3 single-dose injections of EUFLEXXA™ into the target knee; one injection per week at weeks 0, 1 and 2. Patients were followed for 26 weeks following the first injection.
  Interventions: Device: EUFLEXXA™
- Placebo Double-blind (Placebo Comparator): Each subject received 3 single-dose injections of placebo into the target knee; one injection per week at weeks 0, 1 and 2. Patients were followed for 26 weeks following the first injection.
  Interventions: Device: placebo
- EUFLEXXA™ Open Label (Experimental): All patients who participated in the 26 week double-blind study (including participants randomized to the placebo treatment group) and elected to participate in the open label extension, received three injections of EUFLEXXA™ in the target knee. Injections were given once a week on weeks 26, 27 and 28.
  Interventions: Device: EUFLEXXA™

INTERVENTIONS:
Device: EUFLEXXA™ — EUFLEXXA™ is supplied in a single-dose syringe containing 20 mg/2 ml of 1% sodium hyaluronate (molecular weight 2.4-3.6 MD); sodium chloride, 17 mg; disodium hydrogen phosphate dodecahydrate, 1.12 mg; sodium dihydrogen phosphate dihydrate, 0.1 mg; enough water for injection to make 2.0 ml. EUFLEXXA™ is supplied in 2.25 ml nominal volume, disposable prefilled glass syringes containing 2 mL of EUFLEXXA™. Only the contents of the syringe are sterile. EUFLEXXA™ is nonpyrogenic. See package insert for further details.
  Arms: EUFLEXXA™ Double-blind; EUFLEXXA™ Open Label
Device: placebo — Placebo is supplied in a disposable prefilled glass syringe. Each single-dose syringe will contain 2 mL of phosphate buffered saline. Only the contents of the syringe are sterile.
  Arms: Placebo Double-blind

SUMMARY:
This multicenter, randomized, double-blind study will be performed in approximately 600 subjects with chronic idiopathic osteoarthritis (OA) of the knee. An open-label safety extension will follow.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic OA of target knee confirmed by ACR Criteria
2. Pain due to OA in target knee present for at least 6 months:

   • Moderate to severe pain score of 41 mm to 90 mm recorded on a 100 mm VAS immediately following a 50-foot walk
3. A bilateral standing AP X-ray confirming OA of the target knee-obtained within a 6-month period prior to the Screening Visit-and a grade of 2 or 3 according to the Kellgren and Lawrence Grading Scale
4. Ability and willingness to use only acetaminophen as the analgesic (rescue) study medication

   * The acetaminophen dose must not exceed 4 grams/day (4000 mg)
   * If subject has known chronic liver disease, the maximum dose of acetaminophen must not exceed 2 grams/day (2000 mg)
   * The subject must be willing and able to discontinue acetaminophen at least 24 hours prior to all study-specific visits
   * The study specific acetaminophen provided will only be used for knee pain.
5. Ability to perform procedures required of the pain index evaluations (unassisted walking 50 feet on a flat surface and going up and down stairs).
6. Willingness and ability to complete efficacy and safety questionnaires and ability to read and understand study instructions
7. Signed study-specific Subject Informed Consent Form

Exclusion Criteria:

1. Any major injury (including sports injuries) to the target knee within the 12 months prior to the Screening Visit
2. Any surgery to the target knee within the 12 months prior to the Screening Visit, or surgery to the contralateral knee or other weight-bearing joint if it will interfere with knee assessments
3. Prior articular procedures, such as transplants or ligament reconstruction to the target knee
4. Inflammatory arthropathies such as rheumatoid arthritis, lupus arthropathy, or psoriatic arthritis
5. Gout or calcium pyrophosphate (pseudogout) diseases that have flared within the previous 6 months prior to the Screening Visit
6. X-ray findings of acute fractures, severe loss of bone density, avascular necrosis, and/or severe bone or joint deformity in the target knee
7. Osteonecrosis of either knee
8. Fibromyalgia, pes anserine bursitis, lumbar radiculopathy, and/or neurogenic or vascular claudication
9. Significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia in the target knee
10. Significant target knee joint infection or skin disorder/infection within the previous 6 months prior to study enrollment
11. Symptomatic OA of the hips, spine, or ankle, if it would interfere with the evaluation of the target knee
12. Known hypersensitivity to acetaminophen, EUFLEXXA™, or Phosphate buffered saline solution
13. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period
14. Recurrent medical history of severe allergic or immune-mediated reactions or other immune disorders
15. Vascular insufficiency of lower limbs or peripheral neuropathy severe enough to interfere with the study evaluation
16. Current treatment or treatment within the previous 2 years prior to the Screening Visit for any malignancy unless specific written permission is provided by the Sponsor (excluding basal cell or squamous cell carcinoma of the skin)
17. Active liver disease based on liver profile of AST, ALT, and conjugated bilirubin >2 times the upper limit of normal
18. Renal insufficiency based on serum creatinine >2.0 mg/dL
19. Any clinically significant laboratory value based on clinical history that the Investigator feels may affect the study evaluation
20. Any intercurrent chronic disease or condition that may interfere with the completion of the 6-month (or 12-month) follow-up of the study, such as liver disease, severe coronary disease, drug abuse, disordered mental state, or other clinically significant condition
21. Current alcoholism, and/or any known current addiction to pain medications
22. Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study
23. Any psychiatric illness that would prevent comprehension of the details and nature of the study
24. Participation in any experimental drug or device study within the 6 months prior to the Screening Visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site, Los Angeles, California, United States

REFERENCES:
- [Result] Altman RD, Rosen JE, Bloch DA, Hatoum HT. Safety and efficacy of retreatment with a bioengineered hyaluronate for painful osteoarthritis of the knee: results of the open-label Extension Study of the FLEXX Trial. Osteoarthritis Cartilage. 2011 Oct;19(10):1169-75. doi: 10.1016/j.joca.2011.07.001. Epub 2011 Jul 23. PMID 21820521

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 821 patients were screened.
Groups:
- EUFLEXXA™ Double-blind: Each subject received 3 single-dose injections of EUFLEXXA™ (20 milligram/2 milliliter 1 percent sodium hyaluronate) into the target knee; one injection per week at weeks 0, 1 and 2. Patients were followed for 26 weeks following the first injection.
- EUFLEXXA™ Extension Study: Each subject received 3 single-dose injections of EUFLEXXA™ (20 milligram/2 milliliter 1 percent sodium hyaluronate) into the target knee; one injection per week at weeks 26, 27 and 28. Patients were followed for 26 additional weeks (to week 52) following the first injection.
Period: Double-blind
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind | EUFLEXXA™ Extension Study
Started | 293 | 295 | 0
Completed | 257 (Data could not be retrieved for two participants) | 259 (Data could not be retrieved for two participants) | 0
Not Completed | 36 | 36 | 0
Not completed — Adverse Event | 11 | 6 | 0
Not completed — Protocol Violation | 3 | 3 | 0
Not completed — Withdrawal by Subject | 12 | 13 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0
Not completed — Use of exclusionary medication | 1 | 2 | 0
Not completed — Other | 3 | 7 | 0
Not completed — Data could not be retrieved | 2 | 2 | 0
Period: Open-label Extension
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind | EUFLEXXA™ Extension Study
Started | 0 | 0 | 433
Completed | 0 | 0 | 378
Not Completed | 0 | 0 | 55
Not completed — Adverse Event | 0 | 0 | 13
Not completed — Protocol Violation | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 12
Not completed — Use of exclusionary medication | 0 | 0 | 3
Not completed — Other | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind | Total
Number analyzed (Participants) | 293 | 295 | 588
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.62) | 60.8 (10.31) | 61.6 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 186 | 371
  Male | 108 | 109 | 217
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 231 | 228 | 459
  African American | 26 | 33 | 59
  Asian | 5 | 5 | 10
  Hispanic | 29 | 25 | 54
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 293 | 295 | 588
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters square] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to both adult men and women. Body mass index is calculated as weight / (height times height).
  kilograms/meters square | 32.36 (7.446) | 33.03 (7.444) | 32.70 (7.446)
Weight [Mean (Standard Deviation); unit: kilograms] — Mean body weight of study participants in kilograms
  kilograms | 91.0 (21.95) | 92.8 (21.68) | 91.9 (21.81)

OUTCOME MEASURES:

1. Primary Outcome: Observed Pain Scores on 50-foot Walk Test During the Double-blind Study
Description: The level of pain is estimated by the participant following a walk of 50 feet in length which is observed by the investigator. Pain estimates were evaluated on a 100 millimeter visual analog scale. A score of 0 millimeters means there was no pain observed; a score of 100 millimeters means extreme pain was observed.
Time Frame: Weeks 0, 26
Population: Intent to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 291 | 295
units on a scale
  Baseline (Week 0) (n=291,295) | 55.6 (22.06) | 54.7 (21.81)
  Week 26 (n=251,259) | 30.0 (26.06) | 36.1 (28.55)

2. Secondary Outcome: Percent Change From Screening in Observed Pain Scores on 50-foot Walk Test During the Double-blind Study
Description: The percent difference in participant pain recorded by the participant during a walk of 50 feet in length between the screening (week -1) and week 26 scores. Scores are measured on a visual analog scale of 100 millimeters; a score of 0 millimeters means there was no pain observed; a score of 100 millimeters means extreme pain was observed.
Time Frame: weeks -1 and 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percent change from screening value
Arm/Group | EUFLEXXA™ Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 249 | 259
percent change from screening value | -29.3 (277.14) | -38.4 (55.25)
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-Blind vs Placebo Double-Blind; Test type: Superiority or Other; p = 0.008, ANCOVA; Screening pain score was the covariate; study center was modeled as a random effect while all other variables were modeled as fixed effects

3. Secondary Outcome: Percent Change From Baseline in Observed Pain Scores on 50-foot Walk Test During the Double-blind Study for a Subpopulation of Participants With More Severe Knee Pain
Description: Percent difference in participant pain during a walk of 50 feet in length between the mean screening (week -1) and baseline(week 0) scores, and week 26 scores. Scores are recorded by participants and measured on a visual analog scale of 100 millimeters, with 0 millimeters meaning there was no pain observed; 100 millimeters meaning extreme pain was observed.
Time Frame: weeks -1, 0, and 26
Population: Intent to treat population. A subpopulation of patients with more severe knee pain, as measured by having a greater than or equal to 41 millimeter screening score on the 50-foot walk test.
Measure: Mean (Standard Deviation); unit: percentage change from baseline score
Arm/Group | EUFLEXXA™ Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 239 | 254
percentage change from baseline score | -50.5 (42.26) | -36.8 (53.71)
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-Blind vs Placebo Double-Blind; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is purely nominal

4. Secondary Outcome: Number of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the 50-Foot Walk Test at Week 12
Description: Responders are identified based on a calculation of three scales: 50-foot walk test for pain, function and global assessment scales. Each of the individual scales was completed by the participant. A participant was a responder (answer: YES) if there was high improvement in pain or function (>=50 percent and absolute change of >=20 millimeters), or improvement in at least two of three categories: Pain and/or Function and/or Patient Global Assessment scales of >=20 percent and absolute change >=10 millimeter.
Time Frame: Week 12
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 263 | 274
participants
  Yes | 173 | 167
  No | 90 | 107
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.202, Chi-squared

5. Secondary Outcome: Number of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the 50-Foot Walk Test at Week 26
Description: as for outcome 4
Time Frame: Week 26
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 254 | 264
participants
  Yes | 169 | 155
  No | 85 | 109
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.047, Chi-squared

6. Secondary Outcome: Number of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the Western Ontario McMaster University Osteoarthritis Index (WOMAC A) Pain Scale at Week 12
Description: Responders are identified based on a calculation of three scales: WOMAC (A) pain, function and global assessment scales. Each of the individual scales was completed by the participant. A participant was a responder (answer: YES) if there was high improvement in pain or function (>=50 percent and absolute change of >=20 millimeters), or improvement in at least two of three categories: Pain and/or Function and/or Patient Global Assessment scales of >=20 percent and absolute change >=10 millimeter.
Time Frame: Week 12
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 262 | 273
participants
  Yes | 153 | 155
  No | 109 | 118
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.618, Chi-squared

7. Secondary Outcome: Number of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the Western Ontario McMaster University Osteoarthritis Index (WOMAC A) Pain Scale at Week 26
Description: as for outcome 6
Time Frame: week 26
Population: Intent to treat population
Measure: Number; unit: participants
Groups:
- Placebo Double-blind: Each subject received 3 single-dose injections of EUFLEXXA™ into the target knee; one injection per week at weeks 0, 1 and 2. Patients were followed for 26 weeks following the first injection.
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 253 | 264
participants
  Yes | 155 | 137
  No | 98 | 127
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.028, Chi-squared

8. Primary Outcome: Percent Change From Baseline in Observed Pain Scores on 50-foot Walk Test During the Double-blind Study
Description: The percent difference in participant pain recorded by the participant during a walk of 50 feet in length between the baseline (week 0) and week 26 scores. Scores are measured on a visual analog scale of 100 millimeters; a score of 0 millimeters meaning no pain was observed; a score of 100 millimeters meaning extreme pain was observed.
Time Frame: Weeks 0 and 26
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: percent change from baseline value
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 251 | 259
percent change from baseline value | -30.9 (117.20) | -14.9 (114.87)
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.002, ANCOVA; Baseline pain score was the covariate; study center was modeled as a random effect while all other variables were modeled as fixed effects

9. Primary Outcome: Shifts From Extension Study Baseline (Week 26) in Range of Motion Findings at Week 52
Description: Number of participants in various categories of target knee joint examination findings from baseline (week 26 pre-injection) to week 52. Range of motion indicates the flexibility of the knee, and is measured by the number of degrees between when the knee is hyper-extended and when the knee is flexed.
Time Frame: weeks 26 and 52
Population: Safety population which includes all participants who received at least one injection during the extension phase of the study.
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 375
participants
  >135 degrees week 26 / >135 degrees week 52 | 76
  90-135 degrees week 26 / >135 degrees week 52 | 33
  45-89 degrees week 26 / >135 degrees week 52 | 6
  <45 degrees week 26 / >135 degrees week 52 | 0
  >135 degrees week 26 / 90-135 degrees week 52 | 42
  90-135 degrees week 26/ 90-135 degrees week 52 | 171
  45-89 degrees week 26/ 90-135 degrees week 52 | 15
  <45 degrees week 26/ 90-135 degrees week 52 | 2
  >135 degrees week 26 / 45-89 degrees week 52 | 1
  90-135 degrees week 26 / 45-89 degrees week 52 | 12
  45-89 degrees week 26 / 45-89 degrees week 52 | 17
  <45 degrees week 26 / 45-89 degrees week 52 | 0
  >135 degrees week 26 / <45 degrees week 52 | 0
  90-135 degrees week 26 / <45 degrees week 52 | 0
  45-89 degrees week 26 / <45 degrees week 52 | 0
  <45 degrees week 26 / <45 degrees week 52 | 0

10. Primary Outcome: Shifts From Extension Study Baseline (Week 26) in Ratings of Knee Tenderness at Week 52
Description: Number of participants in various categories of target knee joint examination findings from baseline (week 26 pre-injection) to week 52. Tenderness of the knee was subjectively rated by participants as none, mild, moderate or severe.
Time Frame: weeks 26 and 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 377
participants
  None week 26 / none week 52 | 129
  Mild week 26 / none week 52 | 44
  Moderate week 26 / none week 52 | 5
  Severe week 26 / none week 52 | 0
  None week 26 / mild week 52 | 61
  Mild week 26 / mild week 52 | 75
  Moderate week 26 / mild week 52 | 17
  Severe week 26 / mild week 52 | 0
  None week 26 / moderate week 52 | 18
  Mild week 26 / moderate week 52 | 15
  Moderate week 26 / moderate week 52 | 9
  Severe week 26 / moderate week 52 | 1
  None week 26 / severe week 52 | 1
  Mild week 26 / severe week 52 | 1
  Moderate week 26 / severe week 52 | 1
  Severe week 26 / severe week 52 | 0

11. Primary Outcome: Shifts From Extension Study Baseline (Week 26) in Ratings of Knee Local Warmth at Week 52
Description: Number of participants in various categories of target knee joint examination findings from baseline (week 26 pre-injection) to week 52. Local warmth of the target knee was recorded as Yes (warmth present) or No (knee was not warmer than expected).
Time Frame: weeks 26 and 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 377
participants
  Yes week 26 / yes week 52 | 2
  No week 26 / yes week 52 | 11
  Yes week 26 / no week 52 | 11
  No week 26 / no week 52 | 353

12. Primary Outcome: Shifts From Extension Study Baseline (Week 26) in Ratings of Knee Redness at Week 52
Description: Number of participants in various categories of target knee joint examination findings from baseline (week 26 pre-injection) to week 52. Redness of the knee was subjectively rated as Yes (knee was red) and No (knee was not red).
Time Frame: weeks 26 and 52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 377
participants
  Yes week 26 / yes week 52 | 0
  No week 26 / yes week 52 | 0
  Yes week 26 / no week 52 | 4
  No week 26 / no week 52 | 373

13. Secondary Outcome: Change From Baseline in Patient Global Assessment of Knee Pain at Week 26
Description: Participant assessment of knee pain evaluated on a 100 millimeter visual analog scale. A score of 0 millimeters means there was no pain; a score of 100 millimeters means extreme pain.
Time Frame: Weeks 0 and 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 253 | 263
units on a scale | -22.0 (30.38) | -17.8 (28.82)

14. Secondary Outcome: Change From Baseline in the Number of Tablets of Rescue Medication Used at Week 26.
Description: The change in the number of tablets of 500 milligram acetaminophen used in a week as rescue medication is compared at weeks 0 and weeks 26.
Time Frame: Weeks 0 and 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: tablets per week
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 232 | 240
tablets per week | 12.7 (14.56) | 12.9 (15.23)

15. Secondary Outcome: Mean Change From Baseline in Short Form 36 Questionnaire (SF-36) Physical Function (PF) Score at Week 26
Description: The SF-36 questionnaire yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. This table summarizes the change from baseline in participants' physical function. The questionnaire is completed by participants.
Time Frame: Weeks 0, 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EUFLEXXA™ Double Blind: Each subject received 3 single-dose injections of EUFLEXXA™ (20 milligram/2 milliliter 1 percent sodium hyaluronate) into the target knee; one injection per week at weeks 0, 1 and 2. Patients were followed for 26 weeks following the first injection.
Arm/Group | EUFLEXXA™ Double Blind | Placebo Double-Blind
Number analyzed (Participants) | 253 | 264
units on a scale | 4.77 (9.65) | 3.18 (9.05)

16. Secondary Outcome: Mean Change From Baseline in Short Form 36 Questionnaire (SF-36) Bodily Pain(BP) Score at Week 26
Description: The SF-36 questionnaire yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. This table summarizes the change from baseline in participants' bodily pain scores. The questionnaire is completed by participants.
Time Frame: weeks 0 and 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 254 | 265
units on a scale | 3.85 (9.93) | 2.94 (9.56)

17. Secondary Outcome: Mean Change From Baseline in Short Form 36 Questionnaire (SF-36) General Health(GH) Score at Week 26
Description: The SF-36 questionnaire yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. This table summarizes the change from baseline in participants' general health scores. The questionnaire is completed by participants.
Time Frame: weeks 0 and 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 253 | 265
units on a scale | 1.38 (6.22) | 0.19 (6.75)

18. Secondary Outcome: Mean Change From Baseline in Short Form 36 Questionnaire (SF-36) Physical Component Summary (PCS) Score at Week 26
Description: The SF-36 questionnaire yields a score for each domain of health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. The questionnaire is completed by participants. This table summarizes the change from baseline in participants' physical health.
Time Frame: Weeks 0, 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 251 | 263
units on a scale | 4.55 (8.50) | 2.71 (8.58)

19. Secondary Outcome: Number of Participants With 20 Millimeter or Greater Improvement in Pain Scores on the 50-foot Walk Test
Description: Yes represents the number of participants whose pain during a walk of 50 feet in length was improved at week 26 over baseline by at least 20 millimeters. Pain was evaluated on a 100 millimeter visual analog scale by participants. A score of 0 millimeters means there was no pain observed; a score of 100 millimeters means extreme pain was observed.
Time Frame: Weeks 0 and 26
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind
Number analyzed (Participants) | 251 | 259
participants
  Yes | 145 | 120
  No | 106 | 139
Statistical Analysis 1: Comparison: EUFLEXXA™ Double-blind vs Placebo Double-blind; Test type: Superiority or Other; p = 0.006, Chi-squared

20. Secondary Outcome: Observed Pain Scores on the 50-foot Walk Test During the Extension Study
Description: Participant pain during a walk of 50 feet in length was evaluated by participants on a 100 millimeter visual analog scale. A score of 0 millimeters means there was no pain observed; a score of 100 millimeters means extreme pain was observed.
Time Frame: Baseline (week 26), week 52
Population: Intent to treat population. No imputation for missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 425
units on a scale
  Extension baseline (week 26) (n=418) | 33.1 (27.26)
  Week 52 (n=372) | 24.7 (24.88)

21. Secondary Outcome: Mean Change From Baseline in Observed Pain Scores on 50-foot Walk Test During the Extension Study
Description: The mean difference in participant pain as measured by participants during a walk of 50 feet in length between the baseline (week 26 pre-dose) and week 52 scores. Scores are measured on a visual analog scale of 100 millimeters, with a score of 0 millimeters meaning there was no pain observed; a score of 100 millimeters meaning extreme pain was observed.
Time Frame: Extension baseline (week 26), week 52
Population: Intent to treat population. No imputation for missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 367
units on a scale | -7.8 (23.59)

22. Secondary Outcome: Number of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the 50-Foot Walk Test at Week 52
Description: Responders are identified based on a calculation of three scales: 50-foot walk test for pain, function and global assessment scales. Each of the individual scales was completed by the participant. A participant was a responder (answer:YES) if there was high improvement in pain or function (>=50 percent and absolute change of >=20 millimeters), or improvement in at least two of three categories: Pain and/or Function and/or Patient Global Assessment scales of >=20 percent and absolute change >=10 millimeter.
Time Frame: Week 52 (Extension Study)
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 374
participants
  Yes | 144
  No | 230

23. Secondary Outcome: Change From Baseline (Extension Study Week 26) in Use of Rescue Medication at Week 52.
Description: The change in the number of tablets of study-specific acetaminophen taken per week as a rescue medication from knee pain.
Time Frame: Extension baseline (week 26 pre-dose), week 52
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: tablets per week
Arm/Group | EUFLEXXA™ Extension Study
Number analyzed (Participants) | 311
tablets per week | 9.5 (11.90)

ADVERSE EVENTS:
Arm/Group | EUFLEXXA™ Double-blind | Placebo Double-blind | EUFLEXXA™ Extension Study
Serious Adverse Events (participants affected / at risk) | 10/293 | 9/295 | 12/433
Other Adverse Events (participants affected / at risk) | 27/293 | 35/295 | 43/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUFLEXXA™ Double-blind (N=293) | Placebo Double-blind (N=295) | EUFLEXXA™ Extension Study (N=433)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
oophorectomy bilateral (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
bacterial bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUFLEXXA™ Double-blind (N=293) | Placebo Double-blind (N=295) | EUFLEXXA™ Extension Study (N=433)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (27) | 35 (35) | 43 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.